CLINICAL TRIAL: NCT02605902
Title: Randomized Observer Blind Clinical Trial to Demonstrate the Efficacy and Safety of Internet-delivered Behavioral Treatment for Adults With Tic Disorders
Brief Title: Trial to Demonstrate the Efficacy and Safety of Internet-delivered Behavioral Treatment for Adults With Tic Disorders
Acronym: ONLINE-TICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Kirsten Mueller-Vahl, Professor, MD, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: online-tics iCBIT
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2019-10

CONDITIONS: Tics; Tourette Syndrome
Keywords: Chronic tic disorders; Tourette syndrome
MeSH Terms: conditions — Tics; Tourette Syndrome | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- iCBIT (Active Comparator): internet-delivered Comprehensive Behavioral Intervention for Tics (iCBIT) consisting of psychoeducation, habit reversal training (HRT), function-based assessment and intervention, and relaxation training
  Interventions: Behavioral: (i)Comprehensive Behavioral Intervention for Tics
- Control intervention/reference test (Placebo Comparator): internet-delivered psychoeducation and relaxation training.
  Interventions: Behavioral: internet-delivered psychoeducation and relaxation training
- face-to-face CBIT-treatment (Active Comparator): face-to-face CBIT-treatment
  Interventions: Behavioral: (i)Comprehensive Behavioral Intervention for Tics

INTERVENTIONS:
Behavioral: (i)Comprehensive Behavioral Intervention for Tics
  Other Names: (i)CBIT
  Arms: face-to-face CBIT-treatment; iCBIT
Behavioral: internet-delivered psychoeducation and relaxation training
  Arms: Control intervention/reference test

SUMMARY:
Gilles da la Tourette syndrome (TS)* is a common chronic neuropsychiatric disorder characterized by motor and vocal tics. In most adult patients, quality of life is significantly impaired. TS, therefore, is a cost-intensive disease (in Germany: mean total costs=€3404/year). Despite significant adverse effects, dopamine receptor antagonists were recommended as first choice treatment for many years. Although efficacy could be demonstrated only recently, today, behavioral therapy with face-to-face Comprehensive Behavioral Intervention for Tics (CBIT) (including psychoeducation, habit reversal training, function-based assessment and intervention, and relaxation training) is recommended as first line treatment for tics. In Germany, however, dissemination of CBIT is restricted due to a considerable lack of well-trained therapists. The aim of this study is to overcome this deficiency by creating a new and sophisticated internet-delivered CBIT (iCBIT) program. In addition, internet-delivered CBIT will shorten waiting time, will reach additional groups of patients and will be - once developed and established - highly cost-effective (about € 100 vs. € 1450 for face-to-face CBIT). Investigators want to perform a multicenter, randomized, controlled, observer-blind trial including 160 adult patients in order to demonstrate that 8 sessions (10 weeks) of iCBIT are superior to internet-delivered psychoeducation/relaxation in adult patients with TS. Both immediate (1 week after end of treatment) and long-term effects (after 3 and 6 months) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic tic disorder or Tourette syndrome according to DSM-5
* Age ≥18 years; Yale Global Tic Severity Scale (YGTSS) total tic score (TTS) > 14 or > 10 (for patients only with motor or vocal tics)
* Clinical Global Impression-Severity Score (CGI-S) > 4
* Medication for tics and comorbidities must be on a stable dose for at least 6 weeks before entering the study
* Fluent German in speaking and writing
* Ability to give informed consent and signed informed consent

Exclusion Criteria:

* History of schizophrenia or pervasive developmental disorder
* Comorbid obsessive-compulsive disorder (OCD), attention deficit hyperactivity disorder (ADHD), depression, anxiety disorder when unstable and/or in need of an initial adjustment for a therapy
* History of behavioral treatment for tics
* Current illicit substance abuse or addiction (clinically diagnosed)
* Secondary tic disorder or other significant neurological and psychiatric disease
* No internet access or ability to use the internet
* Participation in a study with medicinal products or devices is not allowed within 6 weeks before inclusion or concurrent to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
YGTSS-TTS | 1 week after end of treatment

SECONDARY OUTCOMES:
YGTSS-TTS | 1 week, 3 months and 6 months after end of treatment.
Clinical Global Impression-Improvement Score (CGI-I) | 1 week, 3 months and 6 months after end of treatment.
Clinical Global Impression - Severity Score (CGI-S) | 1 week, 3 months and 6 months after end of treatment.
Modified Rush Video-Based Tic Rating Scale (MRVS) | 1 week, 3 months and 6 months after end of treatment.
Adult Tic Questionnaire (ATQ) (self-report rating) | 1 week, 3 months and 6 months after end of treatment.
Tourette Syndrome-Quality of Life Scale (GTS-QoL) | 1 week, 3 months and 6 months after end of treatment.
Premonitory Urge for Tics Scale (PUTS) | 1 week, 3 months and 6 months after end of treatment.
Beck Depression Inventory (BDI) | 1 week, 3 months and 6 months after end of treatment.
Conners' Adult ADHD Rating Scale (CAARS) | 1 week, 3 months and 6 months after end of treatment.
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 1 week, 3 months and 6 months after end of treatment.
Beck Anxiety Inventory (BAI) | 1 week, 3 months and 6 months after end of treatment.
Working Alliance Inventory-Short Revised (WAI-SR) | 1 week, 3 months and 6 months after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Mueller-Vahl, Prof., MD, Principal Investigator — Medical school Hannover, Clinic for Psychosomatics and Psychotherapy
Locations (5):
- Germany (5):
  - Psychiatric Clinic of the Ludwig-Maximilians-University, Munich, Bavaria
  - Psychotherapist practice, Hanover, Lower Saxony
  - RWTH Aachen, Department of Psychiatry, Psychotherapy and Psychosomatics, Aachen, North Rhine-Westphalia
  - University of Dresden, Dep. of Child and Adolescent Psychiatry, Dresden, Saxony
  - University Medical Center Schleswig-Holstein, UK-SH Campus Lübeck, Department of Neurology, Lübeck, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No